CLINICAL TRIAL: NCT05563363
Title: A Pilot Study on Home Treatment for Individuals Suffering From Severe Addictive Disorders
Brief Title: Home Treatment for Individuals Suffering From Severe Addictive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louise Penzenstadler (Other)
Responsible Party: Sponsor-Investigator, Louise Penzenstadler, Dr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: not yet available
Record Dates: First submitted 2022-09-23; First posted 2022-10-03 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pilot study, randomized, open, non-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home treatment (Experimental): Home visits by care staff at the same frequency as in hospital
  Interventions: Other: Hospital-like treatment in patients' home
- Standard inpatient treatment (Active Comparator): Inpatient treatment on hospital ward
  Interventions: Other: standard inpatient treatment

INTERVENTIONS:
Other: Hospital-like treatment in patients' home — Hospital-like treatment in patients' home. Caregivers, medical doctors and social workers will make several visits per day to the patients' home. 24/7 contact is available.
  Arms: Home treatment
Other: standard inpatient treatment — Inpatient treatment on addiction ward
  Arms: Standard inpatient treatment

SUMMARY:
Home Treatment (HT) has been successfully implemented in adult psychiatry in several countries including Switzerland. Patients with addiction problems were generally excluded even if the latter was not the main diagnosis. On the other hand, community treatments have successfully been established for these individuals. The investigators have recently offered HT to persons with severe addictive disorders which was well accepted.

The investigators intend to conduct a pilot study to prepare a large-scale study if successful. The investigators intend to compare HT to treatment as usual (regular inpatient treatment) on a specialized ward with respect to readmission rates during 6 months after discharge. The data show that 70.8% of all readmissions occur during the first 6 months. Therefore, a period of 6 months is considered an adequate time interval to sufficiently answer this pilot study's question.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder
* age 18 or above
* sufficient french language skills
* competent subjects
* consent to randomization progress

Exclusion Criteria:

* organic brain disease or developmental disorder
* non voluntary admission
* severe somatic comorbidity
* History of complicated substance withdrawal
* acute suicidal ideation
* aggressive behavior
* acute psychiatric disease such as mania or psychosis
* distance to center (must be reachable within 60 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
readmission rates | 6 month post-discharge
  Number of readmissions to hospital during the 6 months following discharge

SECONDARY OUTCOMES:
time to readmission | 6 months
  Number of days between discharge and readmission during the 6 months following discharge
length of hospitalization | 6 months
  total number of days spent in hospital during the 6 months following discharge
number of emergency room visits | 6 months
  number of emergency room visits during the 6 months following discharge
clinical outcome | 6 months
  clinical outcomes measured with Health of the Nation Outcome scale (HoNOS) scoring 0 (no symptoms) to 48 (high symptom level) and the Brief Symptom Check-List (short form of the Brief Symptom Inventory), scoring 0-53 items (higher score = more symptoms). Measured at the start and end of intervention/hospital treatment.
patient satisfaction | 6 months
  Patient satisfaction measured with the S-ANQ (https://www.anq.ch/en/), a questionnaire used by all Swiss hospitals to measure patient satisfaction with treatment. The questionnaire includes 6 questions which are marked from 0 not at all satisfied to 5 = very satisfied. Scoring 0 (not at all satisfied) to 30 (very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No